CLINICAL TRIAL: NCT02068209
Title: Role of Tramadol 50mg in Reducing Pain Associated With Outpatient Hysteroscopy: A Randomized Double Blind Placebo Controlled Trial.
Brief Title: Evaluation of the Role of Tramadol 50mg as an Analgesic During Outpatient Hysteroscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Dr Hassan, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Gany-123
Record Dates: First submitted 2014-02-16; First posted 2014-02-21 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Pain
Keywords: Outpatient hysteroscopy; Tramadol
MeSH Terms: conditions — Pain | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tramadol (Active Comparator): Patients will receive Tramadol 50mg 1 hour before outpatient hysteroscopy
  Interventions: Drug: Tramadol
- Placebo (Placebo Comparator): Patients will receive a placebo 1 hour before the procedure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tramadol — patients will receive Tramadol 50mg orally 1 hour before outpatient hysteroscopy.
  Other Names: Tramadol 50mg
  Arms: Tramadol
Drug: Placebo — patients will receive a placebo 1 hour before outpatient hysteroscopy
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the role of Tramadol 50mg in reducing pain during outpatient hysteroscopy.

DETAILED DESCRIPTION:
This study is a prospective double blinded randomised controlled trial. 140 women will be recruited from the office hysteroscopy clinic in Cairo university hospitals.

All patients attending the outpatient hysteroscopy clinic will be invited to participate in the study. The invitation will include a clear full explanation of the study and patients will provide written consents. Only patients consenting to participate will be included in the trial.

Tramadol and placebo will be enclosed in sealed envelopes which will be numbered using a computer generated random table. Neither the patient nor the physician will be aware of the drug used. Patients will be categorized into 2 groups: Group I who will receive Tramadol 50mg (Tramadol, October Pharma, Giza, Egypt) 1 hour before the procedure, group II who will received a placebo acting as the control group.

Full history will be taken followed by general and local examination. The procedure will be done in the lithotomy position. Hysteroscopy will be done using a 5mm outer diameter continuous flow hysteroscope with a French working channel and a 30 degrees direction of view provided by Techno GmbH and CO. The hysteroscope will be introduced using the vaginoscopy technique, in which no speculum will be used. The cervix will be detected and the external os will be identified using the hysteroscope. The hysteroscope will be introduced in the uterine cavity. Saline will be used as the distension medium and the pressure will be set at 100mm Hg. The anterior wall, posterior wall and tubal ostea will be visualized, any polyps, adhesions septa, congenital malformations or submucous fibroids will be noted.

Base line characteristics will be compared and the main outcome measure will be patients' pain perception during the procedure and 30 minutes later, this will be determined using a visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for outpatient hysteroscopy
* Consent to the procedure

Exclusion Criteria:

* Premenstrual patients
* Known cardiac disease
* Known allergy to Tramadol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Pain perceived by the patient during the procedure | 10 minutes after starting the procedure.
  Pain will be assessed by a visual analogue scale 10 minutes after starting the procedure.

SECONDARY OUTCOMES:
Pain perceived by the patient 30 minutes after the procedure. | 30 minutes after the procedure.
  The level of pain will be assessed 30 minutes after the procedure by a visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: AbdelGany MA Hassan, MRCOG, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

REFERENCES:
- [Background] Floris S, Piras B, Orru M, Silvetti E, Tusconi A, Melis F, Tuveri M, Piga M, Paoletti AM, Melis GB. Efficacy of intravenous tramadol treatment for reducing pain during office diagnostic hysteroscopy. Fertil Steril. 2007 Jan;87(1):147-51. doi: 10.1016/j.fertnstert.2006.05.072. Epub 2006 Nov 1. PMID 17081540
- [Background] Sharma JB, Aruna J, Kumar P, Roy KK, Malhotra N, Kumar S. Comparison of efficacy of oral drotaverine plus mefenamic acid with paracervical block and with intravenous sedation for pain relief during hysteroscopy and endometrial biopsy. Indian J Med Sci. 2009 Jun;63(6):244-52. PMID 19602758
- [Background] van Dongen H, de Kroon CD, Jacobi CE, Trimbos JB, Jansen FW. Diagnostic hysteroscopy in abnormal uterine bleeding: a systematic review and meta-analysis. BJOG. 2007 Jun;114(6):664-75. doi: 10.1111/j.1471-0528.2007.01326.x. PMID 17516956
- [Background] O'Flynn H, Murphy LL, Ahmad G, Watson AJ. Pain relief in outpatient hysteroscopy: a survey of current UK clinical practice. Eur J Obstet Gynecol Reprod Biol. 2011 Jan;154(1):9-15. doi: 10.1016/j.ejogrb.2010.08.015. PMID 20926175
- [Background] Modi H, Mazumdar B, Bhatt J. Study of interaction of tramadol with amlodipine in mice. Indian J Pharmacol. 2013 Jan-Feb;45(1):76-9. doi: 10.4103/0253-7613.106440. PMID 23543914